CLINICAL TRIAL: NCT01224899
Title: Left Cervico-Thoracic Sympathetic Blockade by Clipping in Systolic Heart Failure: A Randomised Controlled Trial
Brief Title: Surgical Sympathetic Blockade in Heart Failure
Acronym: SymBlock
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Paulo Manuel Pego Fernandes, Heart Institute (InCor) HC FMUSP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SymBlock Trial
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Systolic Heart Failure; Beta-blockers Intolerance; Beta-blockers Resistance
Keywords: Heart Failure; Sympathetic Nervous System; Sympathectomy; Adrenergic beta-Antagonists; Ventricular Dysfunction, Left
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Experimental)
  Interventions: Procedure: Left cervico-thoracic sympathetic blockade
- Control (No Intervention)

INTERVENTIONS:
Procedure: Left cervico-thoracic sympathetic blockade — Left cervico-thoracic sympathetic blockade by videothoracoscopic clipping under general anesthesia and single-lumen orotracheal intubation in semi-sitting position.
  Arms: Surgery

SUMMARY:
The investigators sought to evaluate the feasibility and safety of surgical sympathetic blockade in systolic heart failure patients and secondary to assess its cardiovascular consequences.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure (at least 1 month of symptoms onset)
* NYHA functional class II or III
* LV ejection fraction 40% or lower
* resting heart rate higher than 65 bpm
* either maximum beta-blocker therapy according to guidelines or no beta-blocker use for intolerance.

Exclusion Criteria:

* NYHA functional class I or IV
* cardiogenic shock
* resting heart rate ≤ 65 bpm
* systolic blood pressure < 90 mmHg
* sustained ventricular tachycardia
* eligibility to other surgical procedures
* procedure-limiting comorbidity
* presence of ICD or pacemaker
* valvar, chagasic or congenital cardiomyopathy
* age > 70 years
* patient refusal
* contra-indication to videothoracoscopy
* decompensated thyroid disease
* atrial fibrillation or flutter
* active infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Perioperative mortality and morbidity | 30 days after operation
  Study interruption criteria:
  * death attributable to surgical procedure;
  * cardiogenic shock attributable to surgical procedure;
  * worsening of heart failure symptoms attributable to surgical procedure;
  * Horner's syndrome
  * hypotension or bradiarrhythmia attributable to surgical procedure

SECONDARY OUTCOMES:
Cardiovascular effects | 6 months
  * left ventricle ejection fraction (echo and gated blood pool)
  * end left ventricle diastolic diameter
  * mean heart rate
  * heart rate variability
  * New York Heart Association functional class
  * Minesotta Living with Heart Failure Questionnaire Score
  * peak oxygen consumption
  * walked distance in 6 minute walking test
  * BNP
  * 123-I-Metaiodobenzylguanidine (late heart/mediastinum ratio)
  * sympathetic peripheral nerve activity (microneurography)
  * baroreflex parameters (low and high frequency)

CONTACTS AND LOCATIONS:
Overall Officials: Edimar A Bocchi, MD, Study Chair — Heart Institute (InCor) HC FMUSP; Paulo M Pego-Fernandes, MD, Principal Investigator — Heart Institute (InCor) HC FMUSP
Locations (1):
- Heart Institute (InCor) do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Conceicao-Souza GE, Pego-Fernandes PM, Cruz Fd, Guimaraes GV, Bacal F, Vieira ML, Grupi CJ, Giorgi MC, Consolim-Colombo FM, Negrao CE, Rondon MU, Moreira LF, Bocchi EA. Left cardiac sympathetic denervation for treatment of symptomatic systolic heart failure patients: a pilot study. Eur J Heart Fail. 2012 Dec;14(12):1366-73. doi: 10.1093/eurjhf/hfs132. Epub 2012 Oct 25. PMID 23099357